CLINICAL TRIAL: NCT06118398
Title: Effectiveness and Safety of Efgartigimod in the Acute Phase of Neuromyelitis Optica Spectrum Disorders-a Multicentric, Controlled, Retrospective, Real-Word Study
Brief Title: Efgartigimod in Acute Neuromyelitis Optica Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Feng Jinzhou (Other)
Responsible Party: Sponsor-Investigator, Feng Jinzhou, Associate professor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: EANMO-001
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Neuromyelitis Optica; Efgartigimod
MeSH Terms: conditions — Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples are collected before the treatment and at the last visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Intravenous methylprednisolone (IVMP) plus Efgartigimod
  Interventions: Drug: Intravenous methylprednisolone (IVMP) and Efgartigimod
- Control group: IVMP
  Interventions: Drug: IVMP

INTERVENTIONS:
Drug: Intravenous methylprednisolone (IVMP) and Efgartigimod — IVMP 800-1000mg/day for 3-5 days plus Efgartigimod (Efgartigimod: 10mg/kg IV on Day 1, Day 8, Day 15 and Day 22 after IVMP.)
  Groups: Exposed group
Drug: IVMP — IVMP 800-1000mg/day for 3-5 days.
  Groups: Control group

SUMMARY:
This study aims to retrospective investigate the safety and effectiveness of Efgartigimod in the acute phase of neuromyelitis optica spectrum disorders (NMOSD) patients.

DETAILED DESCRIPTION:
This is a multicentre, controlled, retrospective, real-world study which aims to compare the safety and effectiveness of Intravenous methylprednisolone (IVMP) with Efgartigimod injection add-on treatment with IVMP treatment in acute NMOSD patients. Twenty-four patients from 6 centres in China will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years with anti-AQP4-IgG seropositive NMOSD as defined by 2015 NMOSD diagnostic criteria by IPND (International Panel for NMO Diagnosis).
* 2. Patients in the acute phase of NMOSD (definition of acute phase: new neurological symptoms or aggravation of existing symptoms within 30 days before received treatment, lasting at least 24 hours without fever), who had poor response to IVMP and without having received second-line therapies such as plasma exchange or intravenous immunoglobulin consequencely (Poor response is defined as a reduction in EDSS score of: I. <1.0 from the baseline EDSS score when the baseline score was <=5.5 II. < 0.5 when the baseline EDSS score > 5.5).
* 3. Patients who were approved for Efgartigimod treatment would be enrolled in the exposed group.
* 4. Expanded disability status scale (EDSS) score ≤ 8 and ≥ 2.5 before treatment.
* 5. Patients have given their written informed consent.

Exclusion Criteria:

* 1. Lactating and pregnant females before treatment.
* 2. Participated in other interventional studies within 30 days before treatment.
* 3. Received plasma exchange, immunoadsorption, or intravenous immunoglobulin (IVIG） therapy within 1 month before treatment.
* 4. History of malignancies.
* 5. Combined with severe mental disorders and other conditions that unable to cooperate with follow-up.
* 6. After being evaluated by experts, patients with active hepatitis, active tuberculosis, or other special conditions which were ineligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NMOSD patients with acute attacks
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2023-11-05 (Estimated); Primary Completion 2024-11-05 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline. | 1 month
  Change in Expanded Disability Status Scale (EDSS) score from baseline to 1 month after treatment (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Change in Expanded Disability Status Scale (EDSS) score from baseline. | 3 months, 6 months
  Change in Expanded Disability Status Scale (EDSS) score from baseline to 3 months, 6 months after treatment (EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Percentage of Participants with Disability Improvement | 1 month, 3 months, 6 months
  Disability improvement is defined as a reduction in EDSS score of: A) ≥1.0 point from the baseline EDSS score when the baseline score was ≤5.5; B) ≥0.5 point when the baseline EDSS score > 5.5(EDSS: Minimum Score 1, Maximum score 10, higher scores mean a worse outcome).
Change in modified Rankin score (mRS) from baseline. | 1 month, 3 months, 6 months
  Change in modified Rankin score (mRS) from baseline at 1 month 1, 3 month 3 and 6 month (mRS: Minimum Score 0, Maximum score 6, higher scores mean a worse outcome).
Time to first relapse | 6 months
Number of New, and/or Enlarging T2 Hyperintense Lesions Detected by Magnetic Resonance Imaging (MRI) | 6 months
  Number of New, and/or Enlarging T2 Hyperintense Lesions Detected by Magnetic Resonance Imaging (MRI) at the last visit.
Change in timed 25 Foot Walk Test from baseline. | 1 month, 3 months, 6 months
  Change in time taken to complete the timed 25 Foot Walk Test from baseline.
Number of NMOSD attacked during follow-up | 6 months
  Number of NMOSD treatment related to acute attack during follow-up.
Change in serum GFAP levels from baseline | 1 month, 6 months
  Change in serum GFAP levels from baseline to the last visit.
Change in AQP4-ab titres from baseline | 1month, 6 months
  Change in AQP4-ab titres from baseline to the last visit
Change in serum NfL levels from baseline | 1 month, 6 months
  Change in serum NfL levels from baseline to the last visit
Change in Visual Acuity (VA) from baseline | 1 month, 6 months
  Change in Visual Acuity (VA) at1 month 1, and 6 month.
Changes in EQ-5D-5L scores from baseline | 6 months
  Changes in EQ-5D scores from baseline to month 6(EQ-5D-5L: Minimum Score 5, Maximum score 25, lower scores mean a better quality of life).
Change in retinal nerve fibre layer (RNFL) loss from baseline | 1 month,6 months
  Change in retinal nerve fibre layer (RNFL) loss measured by optical coherence tomography (OCT) from baseline at month 1, month 6.
Adverse reactions during treatment and follow-up | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Feng, Ph.D, Principal Investigator — First Affiliated Hospital of Chongqing Medical University

IPD SHARING:
Plan to Share IPD: No